CLINICAL TRIAL: NCT01615393
Title: Prospective, Randomized, Single-blind, Cross-over, Comparative Study for Establishing Comparative Bioavailability of Copegus vs Vilona® in Healthy Volunteers
Brief Title: A Study to Compare the Bioavailability of Copegus and Vilona® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: ML28199
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Ribavirin capsule arm (Active Comparator)
  Interventions: Drug: ribavirin [Vilona]
- Ribavirin tablet arm (Experimental)
  Interventions: Drug: ribavirin [Copegus]

INTERVENTIONS:
Drug: ribavirin [Copegus] — Single oral dose of 400 mg tablets
  Arms: Ribavirin tablet arm
Drug: ribavirin [Vilona] — Single oral dose of a 400 mg capsule
  Arms: Ribavirin capsule arm

SUMMARY:
This prospective, randomized, single-blind, cross-over study will compare the bioavailability of Copegus (ribavirin) administered as tablets and ribavirin administered as capsules in healthy volunteers. Volunteers will be randomized to receive a single dose of 400 mg of ribavirin either as a capsule or as tablets; after a washout phase volunteers will be crossed-over to the other treatment. The anticipated time on study treatment is 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, 18 to 55 years of age
* Clinically healthy as confirmed by medical history, physical examination, electrocardiogram, thorax teleradiography and routine clinical laboratory measurements
* Body mass index between 18 and 28 kg/m2
* Negative testing for drugs of abuse

Exclusion Criteria:

* History or presence of any clinically significant condition that might interfere with the pharmacokinetics of the study drugs
* Volunteers require co-medications during the study
* Exposure to agents known as inducers or inhibitors of hepatic enzymatic system within 30 days prior to study start
* Having taken any medication with a clearance period of over seven half-life before study start
* Hospitalization or significant illness 30 days before study start
* Having received a investigational drug within 90 days prior to study start

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Morelia, Mexico